CLINICAL TRIAL: NCT04643561
Title: A Feasibility Trial Using Trevalan in Healthy Volunteers for Increasing an in Vitro Immune Response to COVID-19 Proteins
Brief Title: Using Travelan to Boost Immune Response in Vitro to COVID-19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Assaf Potruch, MD, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: healthytravelancov19- HMO-CTIL
Record Dates: First submitted 2020-11-24; First posted 2020-11-25 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: hyperimmune colostrum
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): 5 patients will recieve 5 days treatment with Travelan, blood samples will be taken prior and after intervention
  Interventions: Other: Travelan OTC

INTERVENTIONS:
Other: Travelan OTC — 5 days of treatment with Travelan food supplement 3 times a day, blood will be drawn prior and after intervention

SUMMARY:
The gut immune system was shown as an effective target for inducing systemic immune signals against viruses. Oral administration of Travelan, an over the counter product which contains hyperimmune bovine colostrum was shown in preclinical studies to augment the anti-viral immune towards several strains of influenza viruses (RNA viruses).

This study will evaluate the option that Trevalan may help improve the immune system reaction when introduced to COVID-19 proteins in-vitro. 5 healthy volunteers will receive a treatment regimen of 5 days with Trevalan. Before and after treatment, blood samples will be taken in order to test immune response towards viral proteins of the COVID-19 virus in vitro by measuring the number of T cell clone secreting IFNγ against viral antigens.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy volunteers aged 18 years old and above.
2. No history of drug or alcohol abuse.
3. Females of childbearing potential must be non-pregnant (as determined by a serum pregnancy test at screening and again, prior to each dosing session) and agree to use adequate contraceptive means throughout the study.
4. Patients must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.
5. Patients must satisfy a medical examiner about their fitness to participate in the study.
6. Patients must provide written informed consent to participate in the study

Exclusion Criteria:

1. Acute illness resulting in emergency department (ED) evaluation or hospitalization in the last 6 month or any acute illness in the last month before enrollment
2. Patients with evidence of other serious infectious, malignant, autoimmune, kidney, hepatic, or other non-cardiac systemic disease.
3. Chronic drug therapy of any sort
4. Known allergy to milk
5. Over-the-counter drugs, including herbal medications, and prescription drugs (other than those listed above) are not allowed for 4 weeks prior to and throughout the duration of the study
6. Participation in another clinical trial within 30 days prior to intervention.
7. Patients with an inability to communicate well with the PI and staff (i.e., language problem, poor mental development or impaired cerebral function).
8. Patients who will be unavailable for the duration of the trial, are likely to be noncompliant with the protocol, or who are felt to be unsuitable by the PI for any other reason.
9. Known substance abuse, including inhaled or injected drugs in the year prior to Screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
increase levels of IFNγ | 6 days
  The primary objective of this study is to show an increase in levels of IFNγ against viral antigens after treatment regimen with Trevalan

SECONDARY OUTCOMES:
registering adverse events | 30 days
  registering if any adverse events from the use of Travelan

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel